CLINICAL TRIAL: NCT03873532
Title: A Randomized, Open, Multi-center Phase IIb/III Clinical Study to Assess the Efficacy and Safety of Surufatinib Compared to Capecitabine in Advanced or Metastatic Biliary Tract Carcinoma (BTC) Patients
Brief Title: A Trial Evaluating Surufatinib Efficacy and Safety in Biliary Tract Carcinoma Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-012-00CH2
Record Dates: First submitted 2019-03-12; First posted 2019-03-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — surufatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): 300 mg of surufatinib is given by oral administration once a day (QD) every 3 weeks;
  Interventions: Drug: Surufatinib
- Control group (Active Comparator): In each 3-week cycle, Capecitabine is given at 1250 mg/m2 by oral administration twice a day (BID) for 2 weeks, followed by 1 week rest period (equivalent to 2500 mg/m2 total daily dose).
  Interventions: Drug: Capecitabine

INTERVENTIONS:
Drug: Surufatinib — Patients receive oral Surufatinib at a dose of 300mg/d within 1 hour after breakfast (once-daily dosing continuously, every 21-day treatment cycle).
  Other Names: HMPL-012 and Sulfatinib
  Arms: Active group
Drug: Capecitabine — Capecitabine is given at 1250 mg/m2 by oral administration twice a day (BID, one dose each in the morning and evening, with a total dose of 2500 mg/m2 per day) for 2 weeks followed by 1 week of drug interruption. Each course of treatment will last 3 weeks. Capecitabine tablets should be swallowed with water within 30 minutes after a meal.
  Other Names: Xeloda
  Arms: Control group

SUMMARY:
This is a randomized, open-label, active-control, multi-center, phase IIb/III clinical study to evaluate the efficacy and safety of surufatinib vs. Capecitabine as a second-line therapy in patients with unresectable or metastatic biliary tract cancer (BTC). About 298 subjects are randomly assigned to two study treatment groups in the ratio of 1:1 by Interactive Web Response System (IWRS).

* Active group: 300 mg of surufatinib，once a day for 3 weeks as a cycle;
* Control group: In each 3-week cycle, Capecitabine is given at 1250 mg/m2 by oral administration twice a day for 2 weeks, followed by 1 week rest period (equivalent to 2500 mg/m2 total daily dose).

All patients will be treated based on the arm to which they have been randomized. Treatment on study will continue until disease progression, death, intolerable toxicity or other criteria for discontinuation from study treatment. The tumor assessments are performed with imaging every 6 weeks (+3 days) until progressive disease (RECIST v1.1) or death on the study treatment period, and the treatment and survival of the patients after progressive disease are recorded. Safety indicators include adverse events, laboratory tests, vital signs, and changes in electrocardiograms and echocardiograms.

DETAILED DESCRIPTION:
This is a randomized, open-label, active-control, multi-center, phase IIb/III clinical study to evaluate the efficacy and safety of surufatinib vs. Capecitabine as a second-line therapy in patients with unresectable or metastatic biliary tract cancer (BTC). About 298 subjects are randomly assigned to two study treatment groups in the ratio of 1:1 by IWRS.

* Active group: 300 mg of surufatinib is given by oral administration once a day (QD) every 3 weeks;
* Control group: In each 3-week cycle, Capecitabine is given at 1250 mg/m2 by oral administration twice a day (BID) for 2 weeks, followed by 1 week rest period (equivalent to 2500 mg/m2 total daily dose).

Patients are randomized with the following stratification factors:

* Eastern Cooperative Oncology Group (ECOG) Performance Status (0 or 1);
* Years from the first diagnosis of BTC to the randomization date (≤ 1 year or > 1 year);
* The primary site of the tumor (intrahepatic cholangiocarcinoma or extrahepatic cholangiocarcinoma or gallbladder cancer).

All patients will be treated based on the arm to which they have been randomized. Treatment on study will continue until disease progression, death, intolerable toxicity or other criteria for discontinuation from study treatment. The tumor assessments are performed with imaging every 6 weeks (+3 days) until progressive disease (RECIST v1.1) or death on the study treatment period, and the treatment and survival of the patients after progressive disease are recorded. Safety indicators include adverse events, laboratory tests, vital signs, and changes in electrocardiograms and echocardiograms.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are fully informed about the study and voluntarily sign the informed consent (prior to the implementation of any specific procedure for the trial);
2. 18-75 years old (inclusive);
3. Patients with histologically or cytologically confirmed unresectable or metastatic BTC, including intrahepatic cholangiocarcinoma (IHCC), extrahepatic cholangiocarcinoma (EHCC) and gallbladder cancer (GBC);
4. Patients have failed first-line standard systemic chemotherapy. A first-line standard systemic chemotherapy is defined as a regimen of gemcitabine combined with platinum-based therapy. The failure of a first-line standard chemotherapy is defined by progressive disease during the treatment or within 6 months after the last treatment, or intolerable toxicity during the treatment.

   Note: a. The time of first-line medication is ≥ 1 cycle of combination chemotherapy; b. Neoadjuvant or adjuvant chemotherapy is allowed in the early stage, and should be considered failed as a first-line systemic chemotherapy for progressive disease if progressive disease/recurrence occurs during the course of the neoadjuvant/adjuvant therapy or within 6 months after the end of treatment; c. The previous first-line standard chemotherapy does not contain any small molecular anti-angiogenesis agents or monoclonal antibodies, or any drugs related to tumor immunity;
5. ECOG performance status of 0 or 1 (Annex 1);
6. Liver function with a modified Child-Pugh score of < 7;
7. Confirmed measurable (or evaluable) lesions that meet the requirements of RECIST 1.1;
8. Expected survival of ≥ 12 weeks;
9. Fertile male or female patients shall volunteer to use effective contraceptive methods, such as double barrier contraception, condoms, oral or injected contraceptives, and intrauterine devices, during the study period and within 90 days after the last dosing of the investigational drug. All female patients will be considered fertile unless they have had natural menopause, or artificial menopause or sterilization (such as hysterectomy, bilateral adnexectomy or ovarian radiation).

Exclusion Criteria:

1. Received a systemic anti-cancer therapy that has been approved or in development, including chemotherapy, radical radiotherapy, bio-immunotherapy, targeted therapy, and treatment by traditional Chinese medicines (if the instructions of the traditional Chinese medicines specifies clear indications for anti-tumor therapy, the patient may be enrolled after an 1 week of washout period), within 4 weeks prior to randomization;
2. Received a systemic chemotherapy (a neoadjuvant or adjuvant chemotherapy except those that have not failed within 6 months) other than gemcitabine combined with platinum-based therapy (such as fluorouracil-based chemotherapy) prior to randomization; or received an anti-tumor immunotherapy, such as PD-1 and PD-L1 therapies;
3. Received any surgery or invasive treatment/operation (except venous catheterization, puncture and drainage, etc) within 4 weeks prior to randomization;
4. Received any major surgical operations within 60 days before randomization, or have any incisions that have not completely healed;
5. Received a local anti-tumor therapy such as hepatic artery interventional embolization, cryoablation of liver metastases, or radiofrequency ablation within 4 weeks prior to randomization;
6. Patients with any of the following laboratory abnormalities:

   * Absolute neutrophil count (ANC) < 1.5 × 109/L, or platelet (PLT) < 100 × 109/L, or hemoglobin (Hb) < 90 g/L;
   * Total bilirubin ≥ 1.5 × Upper Limit of Normal (ULN);
   * In the absence of liver metastasis, alanine transaminase (ALT) and/or aspartate transaminase (AST) ≥ 1.5 × ULN; in the presence of liver metastasis, ALT and/or AST ≥ 3 × ULN;
   * Serum creatinine ≥ 1.5 × ULN or creatinine clearance < 50 mL/min (calculated according to the Cockcroft-Gault formula, as shown in Annex 2);
   * Routine urinalysis shows urinary protein of ≥ 2+ or 24-hours urinary protein of ≥ 1 g;
7. Uncontrolled malignant ascites (ascites that cannot be controlled by diuretics or puncture as judged by the investigator);
8. Liver metastases accounting for half or more of the total liver volume as determined by the investigator;
9. International normalized ratio (INR) > 1.5 or activated partial thromboplastin time (APTT) > 1.5 × ULN;
10. Clinically significant electrolyte abnormalities as determined by the investigator;
11. Patients with hypertension that is uncontrollable by medications, defined as: systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg;
12. Patients with poorly controlled diabetes mellitus (fasting blood glucose ≥ CTCAE grade 2 after regular treatment);
13. Patients with any disease or condition affecting drug absorption, or patients cannot be treated via oral drug administration;
14. Patients with active gastric and duodenal ulcer, ulcerative colitis and other gastrointestinal diseases, active bleeding caused by unresected tumors, or other conditions that may lead to gastrointestinal bleeding or perforation as judged by the investigator;
15. With evidence or history of apparent bleeding tendency within 3 months prior to randomization (bleeding volume > 30 mL over 3 months, with hematemesis, melena, or hematochezia), hemoptysis (> 5 mL of fresh blood over 4 weeks), or history of thromboembolism within the past 12 months (including stroke and/or transient ischemic attack);
16. With clinically significant cardiovascular diseases, including but not limited to: acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months prior to randomization; congestive heart failure of New York Heart Association (NYHA) grade > 2; ventricular arrhythmias requiring medication; and left ventricular ejection fraction (LVEF) < 50%;
17. Other malignant tumors in the past 5 five years, except basal cell or squamous cell carcinoma that has been treated by radical operation or carcinoma in situ of the cervix;
18. Active or uncontrolled severe infection (≥ CTCAE grade 2) within 2 weeks prior to randomization;
19. Known infection of human immunodeficiency virus (HIV);
20. Known history of clinically significant liver diseases, including viral hepatitis [for known carriers of hepatitis B virus (HBV), the presence of active HBV infection, i.e., positive HBV DNA (> 1 × 104 copies/mL or > 2000 IU/mL), must be excluded; known infection of hepatitis C virus (HCV) with positive HCV RNA (> 1 × 103 copies/mL)], or other hepatitis or cirrhosis;
21. Patients with metastasis in the central nervous system (CNS) or previous brain metastasis;
22. Any unresolved toxicity (> CTCAE grade 1) from previous anti-cancer therapy, excluding alopecia or neurotoxicity of ≤ grade 2 caused by oxaliplatin;
23. Patients participated in clinical trials of other investigational drugs which have not been approved or marketed in China and received corresponding treatment within 4 weeks prior to randomization;
24. Pregnant (positive pregnancy test before dosing) or breast-feeding women;
25. Received transfusion therapy, blood products and hematopoietic factors such as albumin and granulocyte colony stimulating factor (G-CSF) within 14 days prior to randomization;
26. Received brachytherapy (implantation of radioactive particles) within 60 days before the first dose;
27. Any other diseases with clinically significant metabolic abnormalities, abnormal physical observations or abnormal laboratory findings, which are judged by the investigator as evidence that the patient has a disease or condition that is unsuitable for the study drug (e.g., epileptic seizures requiring treatment), or that would interfere with the interpretation of the study results, or that may put the patient at a high risk.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 months after the last patient enrolled.
  Compare the Overall survival (OS) rate between surufatinib group and Capecitabine group.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 5 months after the last patient enrolled.
  Compare the Progression-free survival (PFS) rate between surufatinib group and Capecitabine group.
Objective remission rate (ORR) | 5 months after the last patient enrolled.
  Compare the Objective remission rate (ORR) rate between surufatinib group and Capecitabine group.
Disease control rate (DCR) | 5 months after the last patient enrolled.
  Compare the Disease control rate (DCR) rate between surufatinib group and Capecitabine group.
Duration of response (DOR) | 5 months after the last patient enrolled.
  Compare the Duration of response (DOR) rate between surufatinib group and Capecitabine group.

OTHER OUTCOMES:
Quality of life score | 5 months after the last patient enrolled.
  Compare the Quality of life score between surufatinib group and Capecitabine group. Using quality of life questionnaire (EORTC QLQ-C30) to collect the score. Scale range is 30~126, higher values are considered to be a better outcome.
Changes of tumor markers (CEA, CA199) | 5 months after the last patient enrolled.
  Compare the Changable rate of tumor markers (CEA, CA199) between surufatinib group and Capecitabine group.
Detection of biomarkers | 5 months after the last patient enrolled.
  Correlation between mutation of tumor genes and efficacy; Changes in target-related markers before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rongjun Liu, Study Director — Hutchison Medipharma Limited
Locations (1):
- PLA 307 Hospital, Beijing, Beijing Municipality, China